CLINICAL TRIAL: NCT06362265
Title: A Single Dose Study to Evaluate the Pharmacokinetics of LY3209590 in Pediatric Participants With Type 2 Diabetes Mellitus
Brief Title: A Study to Evaluate Pharmacokinetics of LY3209590 in Pediatric Participants With Type 2 Diabetes Mellitus
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 18437; I8H-MC-BDDB (Other: Eli Lilly and Company)
Record Dates: First submitted 2024-04-09; First posted 2024-04-12 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Insulin
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- LY3209590 (Experimental): LY3209590 administered subcutaneously (SC).
  Interventions: Drug: LY3209590

INTERVENTIONS:
Drug: LY3209590 — Administered SC.

SUMMARY:
The main purpose of this study is to evaluate how much of LY3209590 gets into the blood stream after a single dose and how long it takes the body to remove it in pediatric participants with Type 2 Diabetes Mellitus (T2DM). The study will last for approximately 100 days.

ELIGIBILITY:
Inclusion Criteria:

* Participants with Type 2 Diabetes Mellitus (T2DM) for at least 3 months
* Have Glycated hemoglobin (HbA1c) level of 6.5 percent (%) to 9.5% at screening
* Have a body mass index equal to or less than 45.0 kilograms per square meter (kg/m²)
* Participants are insulin naïve or have been without insulin treatment for at least 3 months prior to screening

Exclusion Criteria:

* Have had a severe hypoglycemia in the past 6 months
* Have a history of renal impairment
* Have had a blood transfusion or severe blood loss within last 90 days
* Have had a significant weight gain or loss of approximately 6% or more within 3 months prior to screening.
* Have a history of an active or untreated malignancy
* Are receiving or received systemic glucocorticoid therapy
* Are currently enrolled in another clinical study trial involving medical research or have participated within the last 30 days in a clinical study involving an investigational product

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Estimated)
Dates: Start 2024-10-10 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetics (PK): Area Under the Plasma Concentration Versus Time Curve (AUC) of LY3209590 | Predose up to 65 days post dose
PK: Maximum Observed Plasma Concentration (Cmax) of LY3209590 | Predose up to 65 days post dose

SECONDARY OUTCOMES:
Change from Baseline in Fasting Glucose | Baseline, 65 days

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (10):
- United States (10):
  - Children's Hospital Los Angeles, Los Angeles, California
  - Children's Healthcare of Atlanta - Center for Advanced Pediatrics, Atlanta, Georgia
  - Centricity Research Columbus Endocrinology, Columbus, Georgia
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Joslin Diabetes Center, Boston, Massachusetts
  - UBMD Pediatrics, Buffalo, New York
  - NYU Langone, New York, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Lifedoc Research - Lenox Park Drive, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://trials.lilly.com/en-US/trial/474857